CLINICAL TRIAL: NCT02588599
Title: A Retrospective Evaluation of the Effect of the Erchonia LUNULA™ on the Increase of Clear Nail in Patients With Toenail Onychomycosis
Brief Title: A Retrospective Analysis of the Effects of Low Level Laser Therapy on Toenail Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_LUNULA_RETRO
Record Dates: First submitted 2015-10-25; First posted 2015-10-28 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia LUNULA (Experimental): The Erchonia LUNULA emits both red light (635 nm) and blue light (405 nm) to the affected toenail for 12 minutes per treatment for 4 treatments, each treatment one week apart.
  Interventions: Device: Erchonia LUNULA

INTERVENTIONS:
Device: Erchonia LUNULA — Active low level laser light therapy

SUMMARY:
The purpose of this study is to determine whether low level laser therapy (LLLT) using the Erchonia LUNULA device is effective in increasing clear nail in toenails with onychomycosis.

DETAILED DESCRIPTION:
Nail onychomycosis, or fungus infection, is typically caused by a fungus called dermatophytes, but may also be caused by yeasts and molds. These microscopic organisms invade the skin through tiny invisible cuts or through a small separation between the nail and the nail bed. Under conditions of warmth and moisture, the fungi grow and spread. The infection begins as a white or yellow spot under the tip of the nail, and as it spreads deeper into the nail, causes unsightly and potentially painful nail discoloration, thickening and the development of crumbling edges. Onychomycosis occurs more commonly in toenails than in fingernails because toenails are often confined in a dark, warm, moist environment inside shoes where fungi can thrive. Toenail fungus affects approximately 23 million people in the US - about 10% of all adults.

Potential complications of onychomycosis include pain in the nails, permanent damage to the nails, development of other serious infections that can spread beyond the feet for individuals with a suppressed immune system due to medication, diabetes or other conditions, such as leukemia and AIDS.

Nail fungus can be difficult to treat, and repeated infections are common. Currently available treatments for onychomycosis include oral antifungal medications, antifungal lacquer, and topical medications, surgical nail removal and photodynamic therapy.

There is no perfect cure for toenail fungus. Even the most effective oral medications are successful only about half of the time, and topical medications are successful less than 10% of the time. Recently, research has found laser therapy to show promise as a novel alternative treatment for toenail onychomycosis. Unlike medication-driven treatments for toenail fungus which can have many side effects including serious ones such as liver toxicity, laser therapy presents minimal to no risk of side effects. Laser therapy is applied to toenail onychomycosis by shining a laser light through the toenail into the tissue below. The laser light vaporizes the fungus while leaving the skin and surrounding healthy tissue unharmed.

Low level laser therapy operates under the principle of photochemistry with a photoacceptor molecule absorbing the emitted photons and inducing a biological cascade. Like our eukaryotic cell, fungi contain the highly complex organelle the mitochondria, which is responsible for the manufacturing of the energy molecule adenosine triphosphate (ATP). Within the inner mitochondrial membrane is cytochrome c oxidase, an identified photoacceptor molecule. It is believed that laser therapy could perhaps provide a means to photo-destroy the fungi responsible for onychomycosis (OM) by inducing the release of highly reactive superoxides. Moreover, laser therapy has been shown to promote superoxide dismutase (SOD), a process responsible for the destruction of foreign invaders. Extracellular release of low levels of mediators associated with SOD can increase the expression of chemokines, cytokines, and endothelial leukocyte adhesion molecules, amplifying the cascade that elicits the inflammatory response. The physiologic function of hydrogen peroxide, superoxide anion, and hydroxyl free radical is to destroy phagocytosed microbes. By enhancing the natural processes of the immune system and impacting the structural integrity of the fungi strain, it is believed that laser therapy may provide a means for clinicians to effectively treat OM without the onset of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Great toenail presents with clearly visually identifiable and photographically documentable onychomycosis of the great toenail, or no visible onychomycosis (1 great toenail)
* Onychomycosis has been identified as due to bacterial/fungal infection classified by the investigator as onychomycosis, with the nail presenting positive on visual inspection for somewhat thickened nail plate with a cloudy appearance and some discoloration (white to yellow to brown)
* Onychomycosis etiology has been confirmed through positive fungal potassium hydroxide preparation (KOH) testing results

Exclusion Criteria:

* Spikes of disease extending to nail matrix in the great toenail
* Infection involving lunula of the great toenail, e.g. genetic nail disorders, primentary disorders
* Great toenail has less than 2mm clear (unaffected) nail plate length beyond the proximal fold
* Dermatophytoma or "yellow spike/streak" (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the great toenail
* Onychogryphosis
* Proximal subungual onychomycosis
* White superficial onychomycosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Zang, DPM, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zang K, Sullivan R, Shanks S. A Retrospective Study of Non-thermal Laser Therapy for the Treatment of Toenail Onychomycosis. J Clin Aesthet Dermatol. 2017 May;10(5):24-30. Epub 2017 May 1. PMID 28670355

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia LUNULA
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) of Toenails Attaining 3 Millimeters (mm) or More of Clear Nail Growth
Description: Individual toenail success criteria was defined as 3 millimeter (mm) or more of clear nail growth at 6 months post-procedure administration as evaluated relative to baseline. Overall study success criteria was defined as an 60% or more of treated toenails meeting the individual success criteria.
Time Frame: 6 Months
Population: Each participant had only one great toenail treated in this study.
Measure: Number; unit: Percent of Toenails
Units Other Than Participants: toenails
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 54
Number analyzed (toenails) | 54
Percent of Toenails | 67

2. Secondary Outcome: Change in Millimeters (mm) of Clear Nail Bed
Description: Millimeter (mm) of clear nail from the base of the toenail was determined from digital photographs of the toenail using a computer program. Change in mm of clear nail bed was calculated as the difference in mm of clear nail bed from baseline measurement to the measurement at 6 months after the end of the procedure administration phase. An increase in mm of clear nail between the two measurement points indicates that the toenail has improved and is positive for study success. A decrease in mm of clear nail between the two measurement points indicates that the toenail has worsened and is negative for study success.
Time Frame: Baseline and 6 Months
Population: Each participant in this study had only one great toenail treated.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: toenails
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 54
Number analyzed (toenails) | 54
millimeters | 5.18 (4.76)
Statistical Analysis 1: Comparison: Erchonia LUNULA; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; t=8.0; df=53

ADVERSE EVENTS:
Arm/Group | Erchonia LUNULA
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No